CLINICAL TRIAL: NCT06381375
Title: Assessment of the Prevalence and the Outcome of Prescribing Drugs Known to Have Major Drug-Drug Interactions With Anti-tuberculous Drugs Among Kasr Alainy Tuberculous Patients
Brief Title: Drug-drug Interactions With Anti-tuberculous Drugs
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Azmy Nabeh, Dr., Cairo University
Other Study IDs: 24-2-2024
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Drug-drug Interaction
MeSH Terms: interventions — Antitubercular Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tuberculous Patients
  Interventions: Other: Anti Tuberculosis Drug

INTERVENTIONS:
Other: Anti Tuberculosis Drug — 1. Estimate the prevalence of prescribing drugs known to have major drug-drug interaction(s) with anti-tuberculous drugs among Kasr Alainy tuberculous patients.
  2. Assess the outcome of prescribing drugs known to have major drug-drug interaction(s) with anti-tuberculous drugs among Kasr Alainy tuberculous patients (response to treatment and the prevalence of life-threatening events).

SUMMARY:
This study aims to assess the prevalence and the outcome of prescribing drugs known to have major drug-drug interactions with anti-tuberculous drugs among Kasr Alainy tuberculous patients.

DETAILED DESCRIPTION:
This study is a longitudinal cohort study that will include all the patients diagnosed with tuberculosis who visit the Tuberculous outpatient clinic at Kasr Alainy after obtaining the approval of the ethical committee, and for about 6 months, to include at least 400 patients as estimated from the sample size calculation result.

A detailed history will be taken including: full name, age, sex( maternity history will be taken in case of female patients to report any current pregnancy or lactation) , mobile number, occupation, history of smoking( cigarette or shisha), type of TB, method of TB diagnosis, history of any comorbidities, current drug(s), and the anti-tuberculous therapy regimen ( including name and dose of each drug), in addition to a baseline liver enzymes( ALT, AST) and a complete blood count (CBC) A written consent will be obtained from the patients, however the study doesn't include any experimental intervention, as it's a pure observational study and it possess no more risk than that encountered in routine daily practice. Patients' confidentiality will be respected and protected. Patients' identity will not be put on the data collection form, and will be replaced by a serial number. This serial study number is linked to the patient identity in a document that will be retained inside the department and will not be used outside the hospital.

Patients will be educated and provided with a sheet (titled drug monitoring diary) to document any drugs that are taken/or will be prescribed concomitantly during the anti-tuberculous therapy in the first month after the initial visit. This diary includes: the drug name, date of start, dose (concentration and frequency), and duration of therapy.

Patients will also be educated and provided with a check list sheet (titled adverse drug events diary, as shown in table 3) to record in a day-by day process any possible adverse drug events for one month, and to score the severity of these events from 1 to 3, as 1 means mild/self-limiting, 2 means moderate/required treatment, 3 severe/life-threatening that needed a specialist consultation and management.

Patients will be educated to deal with expected minor adverse drug events, and will be provided with the contact details of the corresponding researcher who will direct each patient to the corresponding physician accordingly, in case of moderate to severe adverse drug events.

A detailed history of the moderate or severe adverse drug event will be recorded by the researchers, including the (date, symptom(s), and action(s) required to manage that event) Patients are instructed routinely to come for a follow up visit after one month. In this visit, laboratory tests (ALT, AST, CBC) are ordered. The research team will record the laboratory results and the drug monitoring and adverse drug diaries notes. The data will be revised for any missing or conflicting data then the sheets will be prepared for analysis

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with tuberculosis and referred to Tuberculosis outpatient clinic, Kasr Alainy Faculty of Medicine, Cairo University, starting after the obtaining of the Scientific/Ethical approval of the study protocol.

Exclusion Criteria:

* Refusal by the patient/patient's guardian to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with tuberculosis at the tuberculosis outpatient clinic at Kasr Alainy Faculty of Medicine, Cairo University
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Estimate the prevalence of prescribing drugs known to have major drug-drug interaction(s) with anti-tuberculous drugs among Kasr Alainy tuberculous patients | 6 months
2. Assess the outcome of prescribing drugs known to have major drug-drug interaction(s) with anti-tuberculous drugs among Kasr Alainy tuberculous patients (response to treatment and the prevalence of life-threatening events). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Soha Aly Elmorsy, Principal Investigator — Cairo University
Locations (1):
- Omnia Azmy Nabeh, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ghazy RM, Sallam M, Ashmawy R, Elzorkany AM, Reyad OA, Hamdy NA, Khedr H, Mosallam RA. Catastrophic Costs among Tuberculosis-Affected Households in Egypt: Magnitude, Cost Drivers, and Coping Strategies. Int J Environ Res Public Health. 2023 Feb 1;20(3):2640. doi: 10.3390/ijerph20032640. PMID 36768005
- [Background] Yew WW. Clinically significant interactions with drugs used in the treatment of tuberculosis. Drug Saf. 2002;25(2):111-33. doi: 10.2165/00002018-200225020-00005. PMID 11888353